CLINICAL TRIAL: NCT00597922
Title: Variation in Recovery: Role of Gender on Outcomes of Young Acute Myocardial Infarction (AMI) Patients (VIRGO)
Brief Title: Examining Heart Attacks in Young Women
Acronym: VIRGO
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0507000374; R01HL081153-01A1 (NIH)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Heart Attack; Gender Differences; Risk Factors; Quality of Care
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens for biomarker analysis and storage for future genetic studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 2,000 women between the ages of 18 and 55 years who are hospitalized with a heart attack
- 2: 1,000 men between the ages of 18 and 55 years who are hospitalized with a heart attack

SUMMARY:
Heart disease and heart attacks pose a serious health risk to young women, and women tend to experience less successful recoveries after a heart attack than men do. This study will examine various factors that may predispose women to heart attacks and to poor recovery after a heart attack. The differences between men and women in the medical care that they receive following a heart attack will also be studied.

DETAILED DESCRIPTION:
Heart disease is one of the leading causes of death in women 55 years and younger, accounting for more than 8,000 deaths each year in the United States. Approximately 40,000 young women are hospitalized each year in the United States as a result of a heart attack. Research has shown that young women who have heart attacks are twice as likely to die in the hospital as young men who have heart attacks. While there has been an increase in awareness, little research has been conducted on understanding heart disease and heart attacks in young women. Specific biologic markers involved with inflammation, metabolic abnormalities, sex hormones, and genetics may indicate a predisposition to a heart attack and poor recovery. This study will analyze the biologic, demographic, psychosocial, environmental, and behavioral factors that may contribute to premature heart disease and to poor recovery after a heart attack in women. Researchers will examine if delays in receiving medical care following a heart attack can affect recovery and health outcomes for women. Gender differences in outcomes and the quality of medical care that is received following a heart attack will also be examined.

This study will enroll women and men who are hospitalized following a possible heart attack. At study entry, participants will be interviewed to collect information about symptoms, functioning, quality of life, and medical care. A medical record review will also occur. At 1 month after admission from the hospital, an interview will occur via phone and a blood sample will be collected when the participant returns to the hospital or alternatively be collected at a medical clinic convenient to the participant. Another telephone interview will occur at 12 months. Participants' blood samples will be stored for future biologic and genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Elevated cardiac markers within 24 hours of arrival at initial or enrolling institution
* Supporting evidence suggestive of a heart attack

Exclusion Criteria:

* Previously enrolled in the VIRGO study
* Does not speak English or Spanish
* Too ill to interview
* Current prisoner

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 2,000 women and 1,000 men between the ages of 18 and 55 years who are hospitalized with a heart attack
Sampling Method: Non-Probability Sample
Enrollment: 2985 (Actual)
Dates: Start 2007-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harlan M. Krumholz, MD, SM, Principal Investigator — Yale University
Locations (92):
- United States (92):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Sharp Gross Hospital, La Mesa, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center/PRCC Cardiology Research, Los Angeles, California
  - Memorial Medical Center (Sutter Gould Medical Foundation), Modesto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - California Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - St Joseph's Medical Center, Stockton, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Torrance Memorial Medical Center, Torrance, California
  - Denver Health Medical Center, Denver, Colorado
  - Centura Research Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - St Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Hospital of St. Raphael, New Haven, Connecticut
  - Citrus Memorial Health Systems, Inverness, Florida
  - Baptist Cardiac & Vascular Institute, Baptist Hospital of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Pepin Heart Research Institute, Tampa, Florida
  - St Elizabeth's Hospital, Belleville, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Memorial Health System, Springfield, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Krannert Heart Institute - Indiana University - Clarian Methodist Hospital, Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - St Vincent Hospital & Health Services, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Central Maine Heart and Vascular Institute, Lewiston, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St John Hospital & Medical Center, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Mount Clemens Regional Medical Center, Mount Clemens, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St John's Regional Medical Center, Joplin, Missouri
  - Mid-America Heart Institute, St Luke's Hospital, Kansas City, Missouri
  - Heartland Cardiovascular Consultants, Saint Joseph, Missouri
  - Cox South Hospital, Springfield, Missouri
  - St John's Medical Research Institute, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Glacier View Cardiology, Kalispell, Montana
  - The International Heart Institute of Montana, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - The Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Erie County Medical Center, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore/Albert Einstein Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Hospital - Mid Carolina Cardiology, Charlotte, North Carolina
  - Presbysterian Hospital - Mid Carolina Cardiology, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Summa Health System (Akron City Hospital), Akron, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - St Rita's Medical Center, Lima, Ohio
  - Heart Institute of the Cascades, Bend, Oregon
  - Samaritan Heart & Vascular Institute, Corvallis, Oregon
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Clinic - Cardiology, Danville, Pennsylvania
  - Hamot Medical Center, Erie, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - D. Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Sharon Regional Health System, Sharon, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas (UTSW), Dallas, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Sentara Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - St Mary's Medical Center, Huntington, West Virginia
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Derived] Sawano M, Lu Y, Caraballo C, Mahajan S, Dreyer R, Lichtman JH, D'Onofrio G, Spatz E, Khera R, Onuma O, Murugiah K, Spertus JA, Krumholz HM. Sex Difference in Outcomes of Acute Myocardial Infarction in Young Patients. J Am Coll Cardiol. 2023 May 9;81(18):1797-1806. doi: 10.1016/j.jacc.2023.03.383. PMID 37137590
- [Derived] Ding Q, Spatz ES, Lipska KJ, Lin H, Spertus JA, Dreyer RP, Whittemore R, Funk M, Bueno H, Krumholz HM. Newly diagnosed diabetes and outcomes after acute myocardial infarction in young adults. Heart. 2021 Apr;107(8):657-666. doi: 10.1136/heartjnl-2020-317101. Epub 2020 Oct 20. PMID 33082173
- [Derived] Ding Q, Funk M, Spatz ES, Whittemore R, Lin H, Lipska KJ, Dreyer RP, Spertus JA, Krumholz HM. Association of Diabetes Mellitus With Health Status Outcomes in Young Women and Men After Acute Myocardial Infarction: Results From the VIRGO Study. J Am Heart Assoc. 2019 Sep 3;8(17):e010988. doi: 10.1161/JAHA.118.010988. Epub 2019 Aug 23. PMID 31441351
- [Derived] Khera AV, Chaffin M, Zekavat SM, Collins RL, Roselli C, Natarajan P, Lichtman JH, D'Onofrio G, Mattera J, Dreyer R, Spertus JA, Taylor KD, Psaty BM, Rich SS, Post W, Gupta N, Gabriel S, Lander E, Ida Chen YD, Talkowski ME, Rotter JI, Krumholz HM, Kathiresan S. Whole-Genome Sequencing to Characterize Monogenic and Polygenic Contributions in Patients Hospitalized With Early-Onset Myocardial Infarction. Circulation. 2019 Mar 26;139(13):1593-1602. doi: 10.1161/CIRCULATIONAHA.118.035658. PMID 30586733
- [Derived] Safdar B, Spatz ES, Dreyer RP, Beltrame JF, Lichtman JH, Spertus JA, Reynolds HR, Geda M, Bueno H, Dziura JD, Krumholz HM, D'Onofrio G. Presentation, Clinical Profile, and Prognosis of Young Patients With Myocardial Infarction With Nonobstructive Coronary Arteries (MINOCA): Results From the VIRGO Study. J Am Heart Assoc. 2018 Jun 28;7(13):e009174. doi: 10.1161/JAHA.118.009174. PMID 29954744
- [Derived] Lu Y, Ding Q, Xu X, Spatz ES, Dreyer RP, D'Onofrio G, Caulfield M, Nasir K, Spertus JA, Krumholz HM. Sex Differences in Omega-3 and -6 Fatty Acids and Health Status Among Young Adults With Acute Myocardial Infarction: Results From the VIRGO Study. J Am Heart Assoc. 2018 May 30;7(11):e008189. doi: 10.1161/JAHA.117.008189. PMID 29848494
- [Derived] Lu Y, Zhou S, Dreyer RP, Spatz ES, Geda M, Lorenze NP, D'Onofrio G, Lichtman JH, Spertus JA, Ridker PM, Krumholz HM. Sex Differences in Inflammatory Markers and Health Status Among Young Adults With Acute Myocardial Infarction: Results From the VIRGO (Variation in Recovery: Role of Gender on Outcomes of Young Acute Myocardial Infarction Patients) Study. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003470. doi: 10.1161/CIRCOUTCOMES.116.003470. Epub 2017 Feb 22. PMID 28228461
- [Derived] Lindau ST, Abramsohn EM, Bueno H, D'Onofrio G, Lichtman JH, Lorenze NP, Mehta Sanghani R, Spatz ES, Spertus JA, Strait K, Wroblewski K, Zhou S, Krumholz HM. Sexual activity and counseling in the first month after acute myocardial infarction among younger adults in the United States and Spain: a prospective, observational study. Circulation. 2014 Dec 23;130(25):2302-9. doi: 10.1161/CIRCULATIONAHA.114.012709. Epub 2014 Dec 15. PMID 25512442